CLINICAL TRIAL: NCT04712357
Title: Clinical, Control, Double-blind, Randomized Experimentation With Tenofovir Disoproxyl Fumarate and Emtricitabine for COVID-19
Brief Title: Clinical Experimentation With Tenofovir Disoproxyl Fumarate and Emtricitabine for COVID-19
Acronym: ARTAN-C19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Ceara (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); São José Hospital for Infectious Diseases - HSJ (Unknown); Central Laboratory of Public Health of Ceará - Lacen-CE (Unknown)
Responsible Party: Principal Investigator, Aldo Ângelo Moreira Lima, Principal Investigator, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE: 34182620.0.0000.5045
Record Dates: First submitted 2021-01-07; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Covid19
Keywords: Tenofovir; Emtricitabine; COVID-19; Clinical trial
MeSH Terms: conditions — COVID-19 | interventions — Ascorbic Acid; Tablets; Emtricitabine

STUDY DESIGN:
Intervention Model Description: Control case
Who Masked: Participant, Investigator
Masking Description: Randomized double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Vitamin C) (Placebo Comparator): Control placebo (Vitamin C - 500mg / day, for 10 days)
  Interventions: Drug: Vitamin C 500 MG Oral Tablet
- Tenofovir disoproxyl fumarate (TDF) (Active Comparator): Tenofovir disoproxyl fumarate (TDF; 300 mg / day, for 10 days)
  Interventions: Drug: Tenofovir disoproxyl fumarate 300 MG Oral Tablet
- TDF + FTC (Active Comparator): Tenofovir disoproxyl fumarate (TDF; 300 mg / day, for 10 days) plus emtricitabine (FTC; 200 mg / day, for 10 days)
  Interventions: Drug: Tenofovir disoproxyl fumarate 300 MG plus emtricitabine 200 MG Oral Tablet

INTERVENTIONS:
Drug: Vitamin C 500 MG Oral Tablet — Vitamin C 500 MG per day for 10 days
  Arms: Placebo (Vitamin C)
Drug: Tenofovir disoproxyl fumarate 300 MG Oral Tablet — Tenofovir disoproxyl fumarate 300 MG per day for 10 days
  Arms: Tenofovir disoproxyl fumarate (TDF)
Drug: Tenofovir disoproxyl fumarate 300 MG plus emtricitabine 200 MG Oral Tablet — Tenofovir disoproxyl fumarate 300 MG plus emtricitabine 200 MG per day for 10 days
  Arms: TDF + FTC

SUMMARY:
Clinical, control, double-blind, randomized trial with tenofovir disoproxyl fumarate and emtricitabine for Covid-19

DETAILED DESCRIPTION:
Several therapeutic agents have been evaluated for the treatment of Covid-19, and only one using an antiviral drug called remdesivir administered intravenously has shown efficacy to reduce the duration of the disease in 26.7% in critically ill patients. This proposal has as its primary objective (a) Determine the effect of TDF and TDF + FTC on the duration of Covid-19 evaluated in the 14th. day of follow-up at the outpatient clinic in the hospital, duration of the disease observing clinical signs and symptoms, as well as evaluating the RT-PCR viral load tests on the 1st, 7th, 14th. and 28th. days of the study protocol. In addition, the proposal assesses several secondary objectives: (b) Assess the action of TDF and TDF + FTC on the immune response using the rapid ELISA test (IgM / IgG) to be performed on the 7th. and 28th. days of monitoring the experimental protocol; (c) Determine the effect of clinical interventions with the drugs TDF and TDF + FTC in the short and medium term on the viral load of SARS-CoV-2; and (d) Assess the effect of TDF and TDF + FTC on inflammation biomarkers cytokines and chemokines (IL-6, MCP-3, D-dimer, IL1-RA, IL-10, GCSF, TNF-α, MCP-1 , IL-2R, MIP-1 alpha, IP-10, IL-8, NT-proBNP, Troponin I, CRP and procalcitonin) in the blood of patients collected in the 1st, 14th. and 28th. study days. The study will be a prospective, double-blind, placebo control and randomized clinical trial of a total of 219 patients with mild to moderate disease, aged 18 years or over, with clinical signs and symptoms of Covid-19 and certified after the RT-PCR test for the detection of SARS-CoV-2 viral load. The study will be carried out at the outpatient clinic of Hospital São José, Fortaleza, CE. The random groups will be: (1) Group - Placebo control (Vitamin C - 500mg / day, for 10 days); (2) Group - tenofovir disoproxyl fumarate (TDF; 300 mg / day, for 10 days); and (3) Group - TDF + emtricitabine (FTC; 200 mg / day, for 10 days). The study aims to evaluate the efficacy of tenofovir alone or combined with emtricitabine in the duration of mild to moderate Covid-19 cases. The study will also assess the effect of drugs on viral load and immune-inflammatory response. In this sense, the study has the perspective of minimizing the evolution of the disease to severe cases, thus relieving the collapse of the health system and minimizing the social, economic and health disorders of the pandemic by SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 18 years old
* Patient diagnosed with COVID-19

Exclusion Criteria:

* Patient is already receiving some of the study drugs
* There is a hospitalization plan in the next 24h
* Some study treatment is contraindicated
* Patient has HIV infection
* Patient has VHB infection
* Patient lives in another city or state
* Female patient, pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
The time to recovery, defined at day 7 days follow up after enrollment, on which a patient met the criteria for category 1, 2, or 3 on the eight-category ordinal scale. | Day 7 follow up after enrollment.
  The categories are as follows: 1 - No signals and symptoms; 2 - One signal or symptom; 3 - Two signals or symptoms; 4 - Three or more signals or symptoms; 5 - Hospitalized, no active medical problems; 6 - Hospitalized, not on oxygen; 7 - Hospitalized, on oxygen; and 8 - Hospitalized, on high flow oxygen.

SECONDARY OUTCOMES:
SARS-CoV-2 RNA viral load measurements change. | Change between Day 1 and Day 7 follow up after enrollment.
  Molecular diagnostic analyzes will be done by Real-Time PCR (qPCR) based on official guidelines determined by the American CDC (CDC-006-00019, Revision: 03; https://www.fda.gov/media/134922/download). The nasopharyngeal swab samples collected (Covid-19 test) will proceed to the nucleic acid isolation (NuAc). All qPCR reactions will be by uniplex diagnosis. Results will be reported in copies of RNA / mL.
Proportion of patients with qualitative serum IgM / IgG. | Proportion of positive patients at Day 28 for IgM / IgG (N; %).
  The IgM / IgG immune response to SARS-CoV-2 will be qualitative measure using rapid diagnostic test provide by Eco Diagnóstica (Nova Lima, MG, Brazil).
Biomarkers (IL-6, MCP-3, D-dimer, IL1-RA, IL-10, GCSF, TNF-α, MCP-1, IL-2R, MIP-1 alpha, IP-10, IL-8, NT-proBNP, Troponin I, CRP and procalcitonin) measurements change. | Change between Day 1 and Day 14 follow up after enrollment.
  We will use the Luminex XMAP Technology (MAGPIX® System, Merck Co., Kenilworth, NJ) which includes the simultaneous analysis, in the same plasma sample (volume of 25 uL), of a panel of protein markers of pro and anti-inflammatory activity (IL-6, MCP-3, D-dimer, IL1-RA, IL-10, GCSF, TNF-α, MCP-1, IL-2R, MIP-1 alpha, IP-10, IL-8, NT-proBNP, Troponin I). Specific antibodies covalently linked to the carboxylated microspheres containing different specific fluorochromes will be used. Standard curves will be constructed for each protein and then their quantification. Results will be reported in pg / mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Núcleo de Biomedicina - NUBIMED, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No